CLINICAL TRIAL: NCT01288612
Title: Comparative Effectiveness of Endoscopic Assessment of Gastroesophageal Reflux and Barretts Esophagus
Acronym: challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); American College of Gastroenterology (Other)
Responsible Party: Principal Investigator, Prasad G. Iyer, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 10-007787; RC4DK090413 (NIH); UL1TR000135 (NIH)
Record Dates: First submitted 2011-01-28; First posted 2011-02-02 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sedated Endoscopy (Active Comparator): Sedated esophagogastroduodenoscopy with biopsy
  Interventions: Device: Sedated Endoscopy
- Transnasal Endoscopy at Hospital Unit (Active Comparator): Unsedated transnasal endoscopy at hospital unit.
  Interventions: Device: Transnasal Endoscopy
- Transnasal Endoscopy at Mobile Unit (Active Comparator): Unsedated transnasal endoscopy in mobile research van
  Interventions: Device: Transnasal Endoscopy

INTERVENTIONS:
Device: Sedated Endoscopy — The sedated esophagogastroduodenoscopy procedures were performed using a conventional high-definition endoscope (GIF-180, Olympus America, Center Valley, Pennsylvania) under conscious sedation with intravenous midazolam and fentanyl.
  Arms: Sedated Endoscopy
Device: Transnasal Endoscopy — Unsedated transnasal endoscopy performed using the EndoSheath transnasal esophagoscope (TNL-5000, Vision Sciences). Topical anesthetic aerosol spray was applied to the posterior pharynx and nasal spray mixture was applied to the patients nares 10-15 minutes before the endoscopy procedure.
  Arms: Transnasal Endoscopy at Hospital Unit; Transnasal Endoscopy at Mobile Unit

SUMMARY:
The hypothesis of this study was that the comparative effectiveness of unsedated transnasal endoscopy (uTNE) will be greater than sedated endoscopy (sEGD) in population screening for BE.

DETAILED DESCRIPTION:
Barrett's esophagus (BE), a well-known complication of Gastroesophageal Reflux (GER), is the strongest known precursor of esophageal adenocarcinoma. Thus, identifying effective screening approaches for the early detection of BE are highly desired. Current impediments to BE screening include 1) the inability to utilize sedated endoscopy (sEGD) effectively in populations and 2) current GER-based paradigms for detecting BE. Referral center studies demonstrate comparable accuracy between unsedated transnasal endoscopy (uTNE) and sEGD. However, patient acceptability and diagnostic yield with uTNE in general populations remain unknown.

Using the Rochester, Minnesota Epidemiology Project resources, random samples of Olmsted County residents were drawn, and those subjects were mailed validated gastrointestinal symptom questionnaires. These surveys allowed identification of a cohort of community subjects well characterized by the frequency of reflux symptoms. Eligible subjects who were greater than or equal to 50 years old, and who had no previous history of endoscopic evaluation and who were not known to have BE were randomized, stratified by age, sex, and reflux symptoms, and assigned to one of the 3 arms of the study. Subjects in each arm who met the eligibility criteria were initially sent generic invitation letters asking if they agreed to be contacted by phone in two weeks' time to inform them about a research study. If potential subjects explicitly declined to be contacted they were excluded from the study. Eligible subjects were contacted by telephone and only offered the endoscopy technique they had been randomized to. Subjects who accepted and signed an informed consent document were treated according to their randomized assignment and all 3 groups were followed up in the same manner.

Biopsies were taken from any endoscopically suspected BE and from the gastroesophageal junction and squamous mucosa in all subjects. The length of BE segment was defined using Prague criteria. All participants received a telephone call from the research coordinator 1 and 30 days after the procedure to complete validated tolerability scales and adverse events questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Olmsted county, Minnesota resident
* Age 50 or older
* Able to give informed consent

Exclusion Criteria:

* History of known Barretts Esophagus (BE) or endoscopy within the last 10 years
* History of progressive dysphagia
* Known Zenkers or epiphrenic diverticulum
* History of recurrent epistaxis
* Illnesses that impair ability to complete questionnaires (e.g. metastatic cancer, stroke, dementia)
* Contraindication to esophageal biopsy (such as anticoagulation using warfarin or clopidogrel).

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2011-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prasad G. Iyer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Sami SS, Dunagan KT, Johnson ML, Schleck CD, Shah ND, Zinsmeister AR, Wongkeesong LM, Wang KK, Katzka DA, Ragunath K, Iyer PG. A randomized comparative effectiveness trial of novel endoscopic techniques and approaches for Barrett's esophagus screening in the community. Am J Gastroenterol. 2015 Jan;110(1):148-58. doi: 10.1038/ajg.2014.362. Epub 2014 Dec 9. PMID 25488897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were identified using the Rochester Epidemiology Project resources from Olmsted County, Minnesota residents. The study took place between 1 April 2011 and 30 October 2013.
Period: Overall Study
Arm/Group | Sedated Endoscopy | Transnasal Endoscopy at Hospital Unit | Transnasal Endoscopy at Mobile Unit
Started | 150 | 151 | 158
Contacted | 139 | 135 | 138
Agreed to Take Part | 61 | 72 | 76
Completed | 61 | 69 | 76
Not Completed | 89 | 82 | 82
Not completed — Unable to contact | 11 | 16 | 20
Not completed — Declined | 78 | 63 | 62
Not completed — Unable to intubate | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sedated Endoscopy | Transnasal Endoscopy at Hospital Unit | Transnasal Endoscopy at Mobile Unit | Total
Number analyzed (Participants) | 150 | 151 | 158 | 459
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9) | 64 (10) | 64 (10) | 65 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 82 | 87 | 250
  Male | 69 | 69 | 71 | 209
Region of Enrollment [Number; unit: participants]
  United States | 150 | 151 | 158 | 459
Reflux Symptoms [Number; unit: participants]
  Heartburn or acid regurgitation > 1/week | 12 | 16 | 15 | 43
  Heartburn or acid regurgitation < 1/week | 62 | 67 | 68 | 197
  No heartburn or acid regurgitation | 76 | 68 | 75 | 219
Education [Number; unit: participants]
  Less than high school | 2 | 3 | 7 | 12
  High school or some college | 77 | 76 | 72 | 225
  College/professional training | 64 | 67 | 74 | 205
  Unknown/not answered | 7 | 5 | 5 | 17
Employment [Number; unit: participants]
  Employed | 48 | 63 | 56 | 167
  Unemployed/homemaker | 8 | 8 | 11 | 27
  Retired | 87 | 75 | 86 | 248
  Unknown/not answered | 7 | 5 | 5 | 17
Marital Status [Number; unit: participants]
  Married | 115 | 118 | 116 | 349
  Not married (single/widowed/divorced/separated) | 34 | 33 | 41 | 108
  Unknown/not answered | 1 | 0 | 1 | 2
Use of Proton Pump Inhibitor (PPI) [Number; unit: participants]
  Yes | 25 | 23 | 28 | 76
  No | 125 | 128 | 130 | 383

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Agreed to Participated in the Esophageal Assessment
Description: This outcome measure was defined as the proportion of subjects who agreed to undergo esophageal assessment in the three groups out of those who were eligible to be contacted for participation in screening.
Time Frame: Approximately 2 weeks after invitation letter was sent
Population: The analysis population for this outcome measure was the number of subjects per group who were eligible to contact.
Measure: Number; unit: percentage of participants
Arm/Group | Sedated Endoscopy | Transnasal Endoscopy at Hospital Unit | Transnasal Endoscopy at Mobile Unit
Number analyzed (Participants) | 150 | 151 | 158
percentage of participants | 40.7 | 45.7 | 47.5
Statistical Analysis 1: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Mobile Unit; Test type: Superiority or Other; p = 0.25, Chi-squared
Statistical Analysis 2: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Hospital Unit; Test type: Superiority or Other; p = 0.42, Chi-squared
Statistical Analysis 3: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Hospital Unit vs Transnasal Endoscopy at Mobile Unit; Test type: Superiority or Other; p = 0.27, Chi-squared
Statistical Analysis 4: Comparison: Transnasal Endoscopy at Hospital Unit vs Transnasal Endoscopy at Mobile Unit; Test type: Superiority or Other; p = 0.82, Chi-squared

2. Secondary Outcome: Rate of Successful Intubation
Description: The rate of successful intubation was defined as the ability to traverse the upper esophageal sphincter and visualize the esophageal mucosa and classified as successful or unsuccessful.
Time Frame: Visit 1
Population: The analysis population included all subjects who agreed to undergo the esophageal assessment (intent to treat).
Measure: Number; unit: percentage of participants
Arm/Group | Sedated Endoscopy | Transnasal Endoscopy at Hospital Unit | Transnasal Endoscopy at Mobile Unit
Number analyzed (Participants) | 61 | 72 | 76
percentage of participants | 100 | 95.8 | 100
Statistical Analysis 1: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Hospital Unit vs Transnasal Endoscopy at Mobile Unit; Test type: Superiority or Other; p = 0.06, Kruskal-Wallis

3. Secondary Outcome: Rate of Complete Evaluation
Description: The rate of complete evaluation was defined as visualization of the whole esophagus and identification of landmarks: squamocolumnar junction, gastroesophageal junction (upper margin of gastric folds with stomach deflated), and the diaphragmatic hiatus. The categories of evaluation were classified as complete (all three landmarks identified), incomplete (some landmarks identified), or unsuccessful.
Time Frame: Visit 1
Population: The analysis population included all subjects who agreed to undergo the esophageal assessment (intent to treat).
Measure: Number; unit: procedures
Arm/Group | Sedated Endoscopy | Transnasal Endoscopy at Hospital Unit | Transnasal Endoscopy at Mobile Unit
Number analyzed (Participants) | 61 | 72 | 76
procedures
  Complete | 61 | 69 | 75
  Incomplete | 0 | 0 | 1
  Unsuccessful | 0 | 3 | 0
Statistical Analysis 1: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Hospital Unit vs Transnasal Endoscopy at Mobile Unit; Test type: Superiority or Other; p = 0.08, Fisher Exact

4. Secondary Outcome: Rate of Acquisition of Biopsies From the Esophagus
Time Frame: Visit 1
Population: The analysis population included all subjects who agreed to undergo the esophageal assessment (intent to treat).
Measure: Number; unit: percentage of participants
Arm/Group | Sedated Endoscopy | Transnasal Endoscopy at Hospital Unit | Transnasal Endoscopy at Mobile Unit
Number analyzed (Participants) | 61 | 72 | 76
percentage of participants
  Successful | 100 | 83.3 | 79.0
  Unsuccessful | 0 | 16.7 | 21
Statistical Analysis 1: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Hospital Unit vs Transnasal Endoscopy at Mobile Unit; Test type: Superiority or Other; p = 0.001, Kruskal-Wallis

5. Secondary Outcome: Mean Duration of Procedure
Description: Duration of the procedure was defined as time from the beginning of the procedure (initiation of sedation or local anesthesia) to extubation.
Time Frame: Visit 1
Population: The analysis population included all subjects who agreed to undergo the esophageal assessment (intent to treat).
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sedated Endoscopy | Transnasal Endoscopy at Hospital Unit | Transnasal Endoscopy at Mobile Unit
Number analyzed (Participants) | 61 | 72 | 76
minutes | 9.3 (1.6) | 8.0 (2.7) | 8.5 (2.5)
Statistical Analysis 1: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Hospital Unit vs Transnasal Endoscopy at Mobile Unit; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis

6. Secondary Outcome: Mean Time From Extubation to Discharge
Description: This outcome measures the recovery time after the procedure.
Time Frame: Visit 1
Population: The analysis population included all subjects who agreed to undergo the esophageal assessment (intent to treat).
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sedated Endoscopy | Transnasal Endoscopy at Hospital Unit | Transnasal Endoscopy at Mobile Unit
Number analyzed (Participants) | 61 | 72 | 76
minutes | 67.3 (5.9) | 18.5 (4.2) | 15.5 (2.8)
Statistical Analysis 1: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Hospital Unit vs Transnasal Endoscopy at Mobile Unit; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis

7. Secondary Outcome: Mean Tolerability Scores
Description: Validated pain scales (where 0 is none and 10 is severe) were used to assess the degree of pain, choking, gagging, and anxiety experienced during the procedure. Overall tolerance was rated on a scale from 0 to 10, where 0 is good, and 10 is poor tolerance.
Time Frame: Day 1 after the procedure
Population: The analysis population included all subjects who agreed to undergo the esophageal assessment (intent to treat).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sedated Endoscopy | Transnasal Endoscopy at Hospital Unit | Transnasal Endoscopy at Mobile Unit
Number analyzed (Participants) | 61 | 72 | 76
units on a scale
  Pain | 0.1 (0.5) | 2.7 (2.3) | 3.2 (8.8)
  Choking | 0 (0) | 0.8 (1.8) | 0.6 (1.9)
  Gagging | 0.1 (0.6) | 1.2 (2.4) | 1.3 (2.3)
  Anxiety | 0.8 (1.5) | 2.3 (2.2) | 2.8 (2.8)
  Overall Tolerance | 0.4 (0.6) | 2.2 (2.2) | 1.9 (2.2)
Statistical Analysis 1: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Hospital Unit vs Transnasal Endoscopy at Mobile Unit; Comparison between the arms for pain scale; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Hospital Unit vs Transnasal Endoscopy at Mobile Unit; Comparison between the arms for choking scale; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis
Statistical Analysis 3: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Hospital Unit vs Transnasal Endoscopy at Mobile Unit; Comparison between the arms for gagging scale; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Hospital Unit vs Transnasal Endoscopy at Mobile Unit; Comparison between the arms for anxiety scale; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis
Statistical Analysis 5: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Hospital Unit vs Transnasal Endoscopy at Mobile Unit; Comparison between arms for overall tolerance scale; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis

8. Secondary Outcome: Acceptability
Description: Acceptability was defined as the proportion of subjects willing to undergo the procedure again in the future.
Time Frame: Day 1 after the procedure
Population: The analysis population included all subjects who agreed to undergo the esophageal assessment (intent to treat).
Measure: Number; unit: percentage of participants
Arm/Group | Sedated Endoscopy | Transnasal Endoscopy at Hospital Unit | Transnasal Endoscopy at Mobile Unit
Number analyzed (Participants) | 61 | 72 | 76
percentage of participants
  Acceptable | 93.4 | 83.3 | 78.9
  Unacceptable | 6.6 | 16.7 | 21.1
Statistical Analysis 1: Comparison: Sedated Endoscopy vs Transnasal Endoscopy at Hospital Unit vs Transnasal Endoscopy at Mobile Unit; Test type: Superiority or Other; p = 0.001, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 30 days after the procedure
Description: All participants received a telephone call from the research coordinator 1 and 30 days after the procedure to complete adverse events questionnaires.
Arm/Group | Sedated Endoscopy | Transnasal Endoscopy at Hospital Unit | Transnasal Endoscopy at Mobile Unit
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/69 | 0/76
Other Adverse Events (participants affected / at risk) | 14/61 | 20/69 | 23/76
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sedated Endoscopy (N=61) | Transnasal Endoscopy at Hospital Unit (N=69) | Transnasal Endoscopy at Mobile Unit (N=76)
Sore Throat (General disorders) | 8 (8) | 10 (10) | 12 (12)
Bloating (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3)
Epitaxis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) — Self-limiting nose bleed
Nasal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal/chest discomfort (General disorders) | 4 (4) | 4 (4) | 2 (2)
Headache (General disorders) | 0 (0) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes